CLINICAL TRIAL: NCT06953024
Title: Validation of Self Testing Using the INSTI Multiplex HIV1/2 Syphilis Antibody Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Tasha Ramsey, Co-Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 73074
Record Dates: First submitted 2025-04-17; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hiv; Syphilis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Syphilis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- INSTI HIV/syphilis Point of Care Self-Test (Other)
  Interventions: Diagnostic Test: INSTI HIV/syphilis Point of Care Self-Test Administration

INTERVENTIONS:
Diagnostic Test: INSTI HIV/syphilis Point of Care Self-Test Administration — The INSTI Human Immunodeficiency Virus (HIV)/syphilis POCT is a rapid, single-use, flow-through immunoassay that is Health Canada-approved as a screening test for detecting antibodies to HIV1/2 and syphilis using a fingerstick blood sample.

SUMMARY:
This study aims to validate the percent agreement of the INSTI Multiplex Human Immunodeficiency (HIV) 1/2 syphilis antibody (Ab) test (INSTI POCT) when used as a self-test by patients compared to conventional serologic testing.

ELIGIBILITY:
Branch #1: Participants known to have an HIV infection - Inclusion criteria:

• Previously documented positive HIV serology

Branch #2: Participants known to have a history of syphilis infection - Inclusion criteria:

• Documented positive syphilis serology

Branch #3: Participants with no known HIV or syphilis infections - Inclusion criteria:

• No documented positive HIV or syphilis serology

Exclusion criteria:

Unable to speak and understand English

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent agreement of the INSTI HIV/syphilis POCT when used to self-test for antibodies to HIV 1/2 and syphilis when compared to conventional serologic results. | Determined at the end of the implementation period (approximately 6 months).
Participant-rated clarity of instructional materials and satisfaction with INSTI HIV/syphilis self-testing | Immediately after self-testing (Day 0)
  This measure includes two domains assessed immediately following completion of the self-test:
  1. Instructional Clarity: Proportion of participants who agree, are neutral, or disagree with statements related to the clarity and usefulness of the video and infographic
  2. Self-Test Satisfaction: Proportion of participants who agree, are neutral, or disagree with statements related to their satisfaction with the self-testing experience.
  Responses to Likert-style questions will be reported as percentages of participants selecting each category (agree, neutral, disagree) per question.